CLINICAL TRIAL: NCT05962567
Title: Effect of Non-surgical Periodontal Therapy on Interleukin-34 Level in Gingival Crevicular Fluid in Patients With Periodontal Disease (Controlled Clinical Trial)
Brief Title: Interleukin-34 Level in Periodontal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nada Zidan, MSc student, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-Rec IM112108
Record Dates: First submitted 2023-05-12; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Periodontal Disease Stage 2
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Supra and subgingival scaling will be performed on all patients. Oral Hygiene measures will be instructed following treatment and follow up after 3 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy individuals (No Intervention): No intervention
- Stage II periodontitis patients (Active Comparator): Non-surgical periodontal therapy by ultrasonic and universal curettes
  Interventions: Other: Non surgical periodontal therapy

INTERVENTIONS:
Other: Non surgical periodontal therapy — scaling and subgingival debridement
  Arms: Stage II periodontitis patients

SUMMARY:
Aim of the study:

1. To investigate changes in the levels of Interleukin 34 (IL-34) in the Gingival crevicular fluid(GCF) of patients with stage II periodontitis patients before and after nonsurgical periodontal therapy and compare it with healthy individuals
2. To correlate changes in Gingival crevicular fluid level of Interleukin 34 with changes in periodontal parameters after nonsurgical periodontal therapy

DETAILED DESCRIPTION:
Periodontal disease is a chronic disease of various inflammatory diseases where the early symptoms are gingival redness, swelling, and bleeding. As the disease progresses, periodontal pockets, clinical attachment loss (CAL) as well as alveolar bone resorption may occur. If left untreated, periodontal disease can lead to loss of teeth which directly affects patient's mastication.

A new system of periodontal classification has been adopted, in which the types of disease that were previously identified as "chronic" or "aggressive" Armitage, 1999 are now classified under one category ("periodontitis") and re-diagnosed on the basis of many variants (staging and grading system).

The stage is based on the severity of the disease and the complexity of the disease management (in terms of loss of clinical attachment between teeth (CAL), radiographic bone loss, and tooth loss), complexity, and size and distribution. Grading provides additional information about the biological features of the disease, including history-based analysis of the progression rate of periodontitis; progression risk assessment; analysis of possible adverse effects of treatment; and risk assessment that the disease or its treatment may adversely affect the patient's normal life.

Periodontitis is described in four stages ranging from Stage I: Initial periodontitis (CAL 1-2mm), Stage II: Moderate periodontitis (CAL 3-4 mm), Stage III: Severe periodontitis with potential for additional tooth loss (<4), and(CAL≥5mm) Stage IV: Severe periodontitis with potential for loss of dentition (≥5) and (CAL≥5mm). Grading focuses on assessing risk factors like smoking, diabetes, and outcomes of scaling and root debridement. Grade A: Slow rate of progression (no CAL loss over 5 years), Grade B: Moderate rate of progression (CAL loss<2mm over 5years), and Grade C: Rapid rate of progression (CAL loss ≥2 mm over 5 years).

Periodontitis occurs due to a complex of genetic, environmental, and bacterial interaction in which bacterial and host factors play an important role. The imbalance between the previous two factors results in a completely different change from health state to inflammatory disease and once inflammation has begun, activation of many cytokines and molecular mechanisms occur.

Cytokines are defined as soluble small proteins (~5-20 kDa) which bind to specific receptors on certain cells, stimulate some internal cellular changes, and cause multiple genetic and chemical regulations. While molecular mechanisms activate the host-derived proteinase that allow the loss of the marginal periodontal ligament fibers, the migration of the junctional epithelium apically, and the proliferation of bacterial biofilm on the root surface.

There are two different types of inflammatory cytokines: proinflammatory cytokines that is involved in inflammatory reactions including IL-1β, IL-6, IL-12, TNF-α, and anti-inflammatory cytokines that regulate or control the pro-inflammatory cytokine response including IL-4, Interleukin-1 receptor antagonist (IL-1RA) and IL-10

Scaling and root debridement (NSPT) aimed at mechanical removal of bacterial plaque from the tooth surface is considered the "gold standard." This procedure decreases the number of Gram-negative bacteria in favor of Gram-positive bacteria as well as reduces the overall number of microorganisms in periodontal pockets and decrease amount of proinflammatory cytokines.

Traditional clinical periodontal diagnostic parameters used include probing depths, bleeding on probing, clinical attachment levels, plaque index, and radiographs assessing alveolar bone level. They are limited, in that only disease history, not current disease status, can be assessed.

Recent methods in oral and periodontal disease diagnostic research are identifying periodontal risk which is quantified by objective measures like biomarkers which are diagnostic tools to measure periodontal disease at the molecular, cellular, tissue, and clinical levels.

There are many bone resorption biomarkers such as receptor activator nuclear factor kappa B (RANKL), a tumor necrosis factor (TNF) family cytokine, as well as on macrophage colony-stimulating factor (M-CSF) . M-CSF is required for osteoclastogenesis, stimulating both adhesion and proliferation of osteoclast precursors. The novel cytokine interleukin 34 (IL-34) is the second active component of colony-stimulating factor receptor (CSF-1R). IL-34 was shown to stimulate monocyte activation and colonization of macrophages from bone marrow cells.

IL-34 messenger RNA (mRNA) is expressed in a number of tissues, including the heart, brain, lungs, liver, kidneys, spleen, thymus, testes, ovary, small intestine, prostate, and colon, as well as -spleen.

IL-34 plays an important role in RANKL-induced osteoclastogenesis. Inhibition of the CSF-1 receptor by IL-34 has been shown to reduce alveolar bone loss in a periodontal rat model, highlighting their role in periodontal pathology.

The diagnostic potential of gingival crevicular fluid (GCF) has been evaluated from confirming health and disease status to recent predictive tool. It distinguishes between healthy sites of diseased individuals and healthy sites of periodontally healthy people in the microbial profile and the concentration and formation of molecular biomarkers and therefore predicts patient-or-site-based disease Study in 2018, reported that estimation of IL-34 level detects high-risk individuals with periodontitis and systemic diseases, such as diabetes as high levels of IL-34 in gingival crevicular fluid (GCF) and plasma of patients with chronic periodontitis, further increased when accompanied with type 2 diabetes mellitus (T2DM) IL-34 can be considered a potential inflammatory biomarker of periodontal disease as GCF IL-34 levels was high in patients with periodontitis and decreased after NSPT.

On the other hand, salivary levels of IL-34 were significantly lower in the periodontitis group compared to both healthy groups and gingivitis. After receiving non-surgical periodontal treatment at 3 and 6 months post-treatment, IL-34 significantly increased 3 months after treatment compared with baseline.

Therefore, Further studies must be carried out to confirm these findings and to better understand the possible role of IL-34 in the pathogenesis of periodontal diseases and to evaluate its levels in GCF in patients with periodontal disease after non-surgical periodontal treatment (NSPT)

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II Periodontitis.
* Both genders aged from 20-50 years
* Minimum 20 natural teeth excluding third molars
* Good compliance with the plaque control instructions following initial therapy.
* Availability for follow-up and maintenance program.

Exclusion Criteria:

.•Smokers

* Pregnant and lactating females.
* Systemic diseases that could affect the outcome of the therapy (According to Cornell Medical Index-Health Questionnaire).
* Patients taking antibiotics, anti-inflammatory, and immunosuppressive therapy during the preceding 3 months before the start of the trial and during the study.
* Patients who have undergone any periodontal therapy in the last 6 months
* Vulnerable groups of patients e.g. (handicapped patients).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
1- To measure the IL - 34 levels in ng/L in GCF before &after Non-Surgical Periodontal Therapy of stage II periodontitis patients and compare it to healthy individuals | 3 months
  1- To measure the IL - 34 levels in ng/L in GCF before &after Non-Surgical Periodontal Therapy of stage II periodontitis patients and compare it to healthy individuals

SECONDARY OUTCOMES:
To evaluate Plaque index before & after Non-Surgical Periodontal Therapy of stage II periodontitis patients | 3 months
  To evaluate Plaque index (0-3 score) before & after Non-Surgical Periodontal Therapy of stage II periodontitis patients
To evaluate Gingival index before & after Non-Surgical Periodontal Therapy of stage II periodontitis patients | 3 months
  To evaluate Gingival index (0-3 score) before & after Non-Surgical Periodontal Therapy of stage II periodontitis patients
To evaluate Probing depth before & after Non-Surgical Periodontal Therapy of stage II periodontitis patients | 3 months
  To evaluate Probing depth in mm before & after Non-Surgical Periodontal Therapy of stage II periodontitis patients
To evaluate Clinical attachment level before & after Non-Surgical Periodontal Therapy of stage II periodontitis patients | 3 months
  To evaluate Clinical attachment level in mm before & after Non-Surgical Periodontal Therapy of stage II periodontitis patients

CONTACTS AND LOCATIONS:
Overall Officials: Hala A. Abuel Ela, Professor, Study Director — Professor at Faculty of Dentistry, Ain Shams University
Locations (1):
- Faculty of Dentistry-Ain Shams University, Cairo, Egypt

REFERENCES:
- [Result] Dikilitas A, Karaaslan F, Evirgen S, Ertugrul AS. Gingival crevicular fluid CSF-1 and IL-34 levels in patients with stage III grade C periodontitis and uncontrolled type 2 diabetes mellitus. J Periodontal Implant Sci. 2022 Dec;52(6):455-465. doi: 10.5051/jpis.2106260313. Epub 2022 Apr 12. PMID 36468466
- See also: Effect of nonsurgical periodontal therapy on interleukin-34 levels in periodontal health and disease — http://www.ijdr.in/article.asp?issn=0970-9290;year=2018;volume=29;issue=3;spage=280;epage=285;aulast=Guruprasad;type=0